CLINICAL TRIAL: NCT06784388
Title: Clinical Application of Personalized DBS Target Optimization for Treating Depression
Brief Title: Personalized DBS Targeting for Treating Depression
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2024292
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Treatment-resistant Depression (TRD)
Keywords: Treatment-resistant depression (TRD); DBS; stimulation target; stimulation parameters; neural biomarker
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Deep Brain Stimulation; Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Depression (Experimental)
  Interventions: Device: Deep Brain Stimulation(DBS); Drug: Esketamine

INTERVENTIONS:
Device: Deep Brain Stimulation(DBS) — During the DBS treatment phase, the DBS device will apply electrical stimulation to the patient's target brain regions using a specific strategy, and if the efficacy of this phase is not satisfactory, electrical stimulation will continue to be applied during the efficacy observation phase after DBS shutdown.
Drug: Esketamine — SEEG intraoperative experiment: patients will be implanted with microelectrodes and connected to an electrophysiological recorder under local anesthesia. Intraoperative neurophysiological baseline will be recorded for 5 minutes, and esketamine will be injected intravenously at a dose of 0.5 mg/kg, and neurophysiological recordings will be continued for 15 minutes to observe the neuronal electrophysiological changes in various brain regions and target points.

SUMMARY:
The goal of this clinical trial is to optimize the target brain areas for deep brain stimulation (DBS) for depression based on personalized brain imaging and stereo-electroencephalography（SEEG), to administer long-term DBS treatment in the target brain areas, to assess the effectiveness and safety of DBS for refractory depression and to validate the method of personalized optimization of DBS targets. The main questions it aims to answer are:

1. Where is the optimal DBS target brain region for each patient?
2. What are the optimal DBS parameters for each patient ?
3. What are the neural biomarkers of depression symptoms for each patient?
4. Are the optimized DBS strategies effective in treating refractory depression?

DETAILED DESCRIPTION:
This clinical study is a prospective clinical trial focused on the personalized optimization methods and applications of DBS targets for depression.

The study is divided into 4 phases and in each phase and participants will complete different tasks:

1. The preoperative assessment phase:Lasting 7 days, participants will be required to complete preoperative symptom assessments, brain imaging, and task-state functional magnetic resonance imaging(fMRI) assessment.
2. The SEEG assessment phase: Lasting 14 days, participants will be implanted SEEG electrodes and complete a series of SEEG assessments.
3. The DBS treatment phase: Lasting 421 days, participants will be implanted a DBS device and treated with the DBS. During this period, participants will be required to complete the appropriate depressive symptom assessment tasks, as well as follow-up visits every 2 weeks.
4. The efficacy observation phase after DBS shutdown: Lasting 2 months, if the participant has a good outcome at the DBS for depression phase, the electrical stimulation will be shut down for 2 months to observe the maintenance of the efficacy of the treatment, during which time, if the symptoms rebound, the DBS treatment will be restarted until the completion of the study at the end of the 2-month period. During this time participants will be required to complete the appropriate depressive symptom assessment tasks, and follow-up visits every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A psychiatrist-confirmed diagnosis of major depressive disorder in accordance with the Diagnostic And Statistical Manual Of Mental Disorders.5th Ed (DSM-V);
2. A psychiatric examination by two trained psychiatrists and a diagnosis consistent with the DSM-V;
3. A history of depression of at least 12 months duration in depressed patients (including MECT) who have failed to respond to a full dose and course of treatment with 2 or more antidepressants of different mechanisms;
4. A 17-item score on the HAMD scale ⩾ 20 at initial screening;
5. A score of ≤ 50 on the Gross Assessment of Functioning (GAF) scale;
6. The patient himself/herself or legal guardian was able to fully understand the therapy and agreed to enroll after signing an informed consent form.

Exclusion Criteria:

1. Persons with severe or unstable cardiac, hepatic, renal, endocrine, hematologic, and other medical disorders and co-morbidities with psychotic symptoms, including personality disorders diagnosed by history, questioning, and clinical examination;
2. Persons with psychiatric disorders other than depression (except generalized anxiety);
3. Persons with a history of substance abuse within 12 months; persons with a previous history of epilepsy, and persons with febrile convulsions in childhood;
4. Patients with a history of suicide attempts within the past 6 months or more than 2 suicide attempts within the past 2 years;
5. Women who are breastfeeding, pregnant, and patients who are pregnant or intend to become pregnant during the clinical study;
6. Contraindications to DBS surgery and MRI;
7. Years of education less than or equal to 9 years;
8. Patients who are involuntarily hospitalized.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Rating Scale for Depression (HAMD) score during the DBS treatment phase relative to preoperative baseline | at baseline and after 442 day
  Improvement is defined as a 25-49% reduction in Hamilton Rating Scale for Depression (HAMD) score relative to the preoperative baseline; response is defined as a ≥50% reduction in HAMD score relative to the preoperative baseline; and remission is defined as a HAMD score ≤8.
Changes in HAMD scores during the efficacy observation phase after DBS shutdown | Two months after 442 days
  Rebound is defined as a HAMD ≥18 in the subsequent follow-up period if the patient has an initial assessment of HAMD ≤8 in the efficacy observation phase after DBS shutdown, and rebound is defined as a HAMD score more than 2 times the initial assessment or 20 in the subsequent follow-up period if the patient has an initial assessment of HAMD >8 in that phase.

SECONDARY OUTCOMES:
the score of Montgomery-Asberg Depression Rating Scale (MADRS) | Every 2 weeks between day 21 and day 442
  The score of the scale ranges from 0 to 60. Higher MADRS score indicates more severe depression.
the score of multi-lingual Hypomania Check List(C-SSRS) | Every 2 weeks between day 21 and day 442
  The Multi-Lingual Hypomania Check List (C-SSRS) is a self-report questionnaire used to assess hypomanic symptoms and suicide risk. This tool includes multiple items designed to identify emotional and behavioral changes based on patient feedback. The results of the C-SSRS assist professionals in developing treatment plans, with higher scores typically indicating more severe symptoms, thereby facilitating timely intervention and support.
the score of Hamilton Anxiety Scale(HAMA) | Every 2 weeks between day 21 and day 442
  The score of the scale ranges from 0 to 56. The higher scores means more severe anxiety.
the score of the Oxford Depression Questionnaire(ODQ) | Every 2 weeks between day 21 and day 442
  The Oxford Depression Questionnaire (ODQ) is a self-report instrument designed to assess the presence and severity of depressive symptoms. It evaluates various aspects of mood, motivation, and behavior related to depression. The questionnaire consists of multiple items scored on a scale, where higher scores indicate greater levels of depressive symptoms, facilitating effective monitoring and intervention by healthcare professionals.
the score of THINC-integrated tool(THINC-it) | Every 2 weeks between day 21 and day 442
  Neuropsychological measures contains six domains of cognition which are episodic memory, working memory,attention, executive functions, psychomotor speed and social cognition.
the score of Visual Analogue Scale-Depression(VAS-D) | Every 2 weeks between day 21 and day 442
  The Visual Analogue Scale for Depression (VAS-D) is a self-report tool used to assess the severity of depressive symptoms. It consists of a single continuous line, where respondents indicate their level of depression by marking a point on the line. The scale ranges from "no depression" to "worst possible depression," allowing for a visual representation of the individual's emotional state. Higher marks on the scale correspond to greater levels of depressive symptoms, aiding healthcare providers in monitoring and addressing the patient's condition.
the score of HAMD-6 item(HAMD-6) | Every 2 weeks between day 21 and day 442
  The Hamilton Depression Rating Scale-6 Item (HAMD-6) is a self-report questionnaire designed to assess the severity of depression. It focuses on six key symptoms, including mood, feelings of guilt, insomnia, work and activities, psychomotor agitation or retardation, and anxiety. Each item is rated on a scale, with higher scores indicating more severe depressive symptoms. This concise tool facilitates quick evaluation and monitoring of depression in clinical settings.
the score of Patient Health Questionnaire-9( PHQ-9) | Every 2 weeks between day 21 and day 442
  The Patient Health Questionnaire-9 (PHQ-9) is a self-report tool used to assess the presence and severity of depressive symptoms. It consists of nine items that correspond to the diagnostic criteria for major depressive disorder. Respondents rate the frequency of their symptoms over the past two weeks on a 4-point scale. Higher scores indicate more severe depressive symptoms, helping healthcare providers to evaluate, monitor, and guide treatment decisions for patients.
the score of Beck Depression Inventory(BDI) | Every 2 weeks between day 21 and day 442
  The Beck Depression Inventory (BDI) is a self-report questionnaire designed to measure the severity of depressive symptoms. It consists of 21 items that assess various aspects of depression, including mood, hopelessness, and physical symptoms. Respondents rate each item on a scale, with higher scores indicating greater levels of depression. The BDI is widely used in clinical and research settings to evaluate depression and monitor treatment progress.
the score of Visual Analogue Scale-Anxiety(VAS-A) | Every 2 weeks between day 21 and day 442
  The Visual Analogue Scale for Anxiety (VAS-A) is a self-report tool used to measure the level of anxiety experienced by individuals. It consists of a continuous line, where respondents indicate their anxiety level by marking a point on the line. The scale ranges from "no anxiety" to "worst possible anxiety," providing a visual representation of the individual's emotional state. Higher marks on the scale correspond to greater levels of anxiety, assisting healthcare providers in assessing and addressing the patient's anxiety levels.
the score of General Anxiety Disorder-7(GAD-7) | Every 2 weeks between day 21 and day 442
  The Generalized Anxiety Disorder-7 (GAD-7) is a self-report questionnaire designed to assess the severity of generalized anxiety disorder symptoms. It consists of seven items that evaluate various aspects of anxiety, including feelings of nervousness, worry, and difficulty relaxing. Respondents rate the frequency of their symptoms over the past two weeks on a 4-point scale. Higher scores indicate more severe anxiety symptoms, helping healthcare providers to identify and monitor anxiety levels in patients effectively.
the score of Beck Anxiety Inventory(BAI) | Every 2 weeks between day 21 and day 442
  The Beck Anxiety Inventory (BAI) is a self-report questionnaire designed to measure the severity of anxiety symptoms. It consists of 21 items that assess various aspects of anxiety, such as physiological symptoms and cognitive disturbances. Respondents rate the intensity of their anxiety over the past week on a 4-point scale. Higher scores indicate greater levels of anxiety, providing valuable information for healthcare providers in evaluating and managing anxiety disorders.
the score of Immediate Mood Scale(IMS) | Every 2 weeks between day 21 and day 442
  The Immediate Mood Scale (IMS) is a self-report questionnaire designed to assess an individual's current mood state. It includes a series of items that evaluate various emotional dimensions, such as happiness, sadness, anxiety, and anger. Respondents rate their mood on a scale, providing a snapshot of their emotional well-being at the moment. Higher scores on specific mood dimensions indicate a more positive emotional state, assisting healthcare providers in understanding and addressing the individual's immediate emotional needs.
the score of Quick Inventory of Depressive Symptomatology, Self-Rated(QIDS-SR) | Every 2 weeks between day 21 and day 442
  The score of the scale ranges from 0 to 42. Higher QIDS-SR16 score indicates more severe depression.
Adverse events | Perioperative and every 2 weeks between day 21 and day 442
  Record: Adverse events during the "perioperative period" of SEEG and DBS implantation, during the DBS treatment phase, and during the follow-up period of the efficacy observation phase after DBS shutdown , including abnormalities in laboratory tests as judged necessary by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scangos KW, Khambhati AN, Daly PM, Makhoul GS, Sugrue LP, Zamanian H, Liu TX, Rao VR, Sellers KK, Dawes HE, Starr PA, Krystal AD, Chang EF. Closed-loop neuromodulation in an individual with treatment-resistant depression. Nat Med. 2021 Oct;27(10):1696-1700. doi: 10.1038/s41591-021-01480-w. Epub 2021 Oct 4. PMID 34608328
- [Background] Alagapan S, Choi KS, Heisig S, Riva-Posse P, Crowell A, Tiruvadi V, Obatusin M, Veerakumar A, Waters AC, Gross RE, Quinn S, Denison L, O'Shaughnessy M, Connor M, Canal G, Cha J, Hershenberg R, Nauvel T, Isbaine F, Afzal MF, Figee M, Kopell BH, Butera R, Mayberg HS, Rozell CJ. Cingulate dynamics track depression recovery with deep brain stimulation. Nature. 2023 Oct;622(7981):130-138. doi: 10.1038/s41586-023-06541-3. Epub 2023 Sep 20. PMID 37730990